CLINICAL TRIAL: NCT00322335
Title: Phase III, Open, Multicenter Study to Assess the Long-Term Persistence of a Booster Dose of GSK Biologicals' Hib-MenC Compared to a Booster Dose of Infanrix™ Hexa When Given to 14 Month-old Subjects Primed in Study DTPa-HBV-IPV-097 & Boosted in Study Hib-MenC-TT-010 BST: DTPa-HBV-IPV-097
Brief Title: Long-term Persistence Study to Assess a Booster Dose of GSK Biologicals' Hib-MenC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106672; 106673 (Other: GSK); 106675 (Other: GSK); 106679 (Other: GSK); 106680 (Other: GSK)
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: H.influenzae type b Disease
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines; Engerix-B

ARMS (3):
- Menitorix/Pediarix Group (Experimental): Subjects were primed with 3 doses of Pediarix™ co-administered intramuscularly with Menitorix™ in the right and left thigh respectively in the primary study (NCT00352963) at 2, 4 and 6 months of age. This was followed by a booster dose of Menitorix™ administered intramuscularly in the left thigh between 13 and 14 months of age in study NCT00323050. No vaccines were administered during this long-term persistence phase of the study.
  Interventions: Biological: Haemophilus influenzae type b- and meningococcal (vaccine); Biological: Infanrix™ penta
- Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group (Active Comparator): Subjects were either primed in the primary study (NCT00352963) with 3 doses of Infanrix™ hexa administered intramuscularly in the right thigh at 2, 4 and 6 months of age and 2 doses of NeisVac-C™ administered intramuscularly in the left thigh at 2 and 4 months of age or with Engerix-B at birth intramuscularly in the right thigh, Infanrix™ hexa intramusculary in the right thigh at 2 and 6 months of age and NeisVac-C™ intramuscularly in the left thigh at 2 and 4 months of age, Infanrix™ IPV/Hib was administered intramuscularly in the right thigh at 4 months of age. All subjects were boosted with Menitorix™ administered intramuscularly in the left thigh between 13 and 14 months of age in study NCT00323050. No vaccines were administered during this long-term persistence phase of the study.
  Interventions: Biological: Haemophilus influenzae type b- and meningococcal (vaccine); Biological: Infanrix™ hexa; Biological: Engerix-B; Biological: NeisVac-C™; Biological: Infanrix™ IPV/HIB
- Infanrix hexa/Meningitec Group (Active Comparator): Subjects were primed with Infanrix™ hexa co-administered intramuscularly with Meningitec™ in the right and left thigh respectively at 2, 4 and 6 months of age during the primary study (NCT00352963), followed by a booster dose of Infanrix™ hexa intramuscularly in the right thigh between 13 and 14 months of age in study (NCT00323050). No vaccines were administered during this long-term persistence phase of the study.
  Interventions: Biological: Infanrix™ hexa; Biological: Meningitec™

INTERVENTIONS:
Biological: Haemophilus influenzae type b- and meningococcal (vaccine) — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age (group HibMenC) and as booster dose at 14 months of age (groups HibMenC and group NeisPoo).
  Arms: Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group; Menitorix/Pediarix Group
Biological: Infanrix™ penta — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age
  Arms: Menitorix/Pediarix Group
Biological: Infanrix™ hexa — Intramuscular injection into the thigh as primary vaccination at 2, 4 and/or 6 months of age (groups NeisPoo and MenCCRM) and/or as booster dose at 14 months of age (group MenCCRM).
  Arms: Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group; Infanrix hexa/Meningitec Group
Biological: Engerix-B — Intramuscular injection into the thigh as a birth dose
  Arms: Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group
Biological: NeisVac-C™ — Intramuscular injection into the thigh as primary vaccination at 2 and 4 months of age.
  Arms: Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group
Biological: Infanrix™ IPV/HIB — Intramuscular injection into the thigh as primary vaccination at 4 months of age
  Arms: Infanrix hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group
Biological: Meningitec™ — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age
  Arms: Infanrix hexa/Meningitec Group

SUMMARY:
This protocol posting deals with objectives & outcome measures of the extension phase at Months 18, 30, 42, 54 and 66 post booster. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00352963). The objectives & outcome measures of the Booster phase/study are presented in a separate protocol posting (NCT number =NCT00323050).

The purpose of this study is to evaluate the persistence of meningococcal serogroup C and Hib antibodies on a yearly basis for a period of 5.5 years after booster vaccination. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This multicenter study is open. No vaccine will be administered during this persistence phase of the study. The subjects were randomized in the primary vaccination study 217744/097 (DTPa-HBV-IPV-097) and will not be further randomized in this study. The study has 3 groups with Meningitec™ primed group as control. The protocol was amended to allow for enrollment of subjects of the Meningitec™ primed control group who were boosted with Meningitec™ after the end of the booster study as per new local reccommendation in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female in their third year of life at the time of the study initiation for the subjects who enter the study at Visit 1. The subjects who enter the study at Visit 2 should be in their fourth year of life at the time of the study initiation.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having completed the booster vaccination study Hib-MenC-TT-010 BST:DTPA-HBV-IPV-097 (NCT=00323050).
* Subjects who are part of the Meningitec™ control group and who were not enrolled at Visit 1 can be enrolled at Visit 2 if they have completed the booster vaccination study Hib-MenC-TT-010 BST:DTPA-HBV-IPV-097 (NCT=00323050) and if they have received a fourth dose of Meningitec™ in their second year of life, after the booster study Hib-MenC-TT-010 BST:DTPA-HBV-IPV-097 (NCT=00323050)

Exclusion Criteria:

* Previous administration of a booster dose of Hib or meningococcal serogroup C except booster study vaccines during the study Hib-MenC-TT-010 BST:DTPA-HBV-IPV-097. Subjects who received a 4th dose of Meningitec™ should be included in the study.
* History of H. influenzae type b, meningococcal serogroup C diseases.

Ages: 31 Months to 33 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Spain (10):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vélez-Málaga / Málaga

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Tejedor JC, Moro M, Merino JM, Gomez-Campdera JA, Garcia-del-Rio M, Jurado A, Diez-Delgado FJ, Omenaca F, Garcia-Sicilia J, Ruiz-Contreras J, Martin-Ancel A, Roca J, Boceta R, Garcia-Corbeira P, Maechler G, Boutriau D; Spanish 102547 Study Group. Immunogenicity and reactogenicity of a booster dose of a novel combined Haemophilus influenzae type b-Neisseria meningitidis serogroup C-tetanus toxoid conjugate vaccine given to toddlers of 13-14 months of age with antibody persistence up to 31 months of age. Pediatr Infect Dis J. 2008 Jul;27(7):579-88. doi: 10.1097/INF.0b013e31816b4561. PMID 18536619
- [Background] Tejedor JC, Merino JM, Moro M, Navarro ML, Espin J, Omenaca F, Garcia-Sicilia J, Moreno-Perez D, Ruiz-Contreras J, Centeno F, Barrio F, Cabanillas L, Muro M, Esporrin C, De Torres MJ, Caubet M, Boutriau D, Miller JM, Mesaros N. Five-year antibody persistence and safety following a booster dose of combined Haemophilus influenzae type b-Neisseria meningitidis serogroup C-tetanus toxoid conjugate vaccine. Pediatr Infect Dis J. 2012 Oct;31(10):1074-7. doi: 10.1097/INF.0b013e318269433a. PMID 22828645
- [Background] Tejedor JC et al. Antibody persistence 54 months after a booster dose of combined Haemophilus influenzae type b-Neisseria meningitidis serogroup C-tetanus-toxoid (HibMenC-TT) conjugate vaccine. Abstract presented at the 29th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID). The Hague, The Netherlands, 7-11 June 2011.
- [Background] Tejedor JC et al. Antibody persistence 66 months after a booster dose of combined Haemophilus influenzae type B-Neisseria meningitidis serogroup C-tetanus-toxoid (Hib-MenC-TT) conjugate vaccine. Abstract presented at the 30th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID), Thessaloniki, Greece, 8-12 May 2012.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 106672 are summarised with studies 106673, 106675, 106679, and 106680 on the GSK Clinical Study Register.
- Available data/document: Clinical Study Report: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106672 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The follow-up timepoints include all subjects who came back for that timepoint. Therefore the amount of subjects who completed the previous timepoint does not correspond with the amount of subjects starting the following time-point per se.
Period: Subjects 18 Months After Booster Dose
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Started | 58 | 123 | 3 (Subjects who received Meningitec booster outside scope study NCT00323050 eliminated from this period)
Completed | 58 | 123 | 3
Not Completed | 0 | 0 | 0
Period: Subjects 30 Months After Booster Dose
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Started | 54 | 119 | 57 (Subjects eliminated from previous timepoint were included again from this timepoint onwards)
Completed | 54 | 119 | 57
Not Completed | 0 | 0 | 0
Period: Subjects 42 Months After Booster Dose
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Started | 51 | 113 | 56
Completed | 51 | 113 | 56
Not Completed | 0 | 0 | 0
Period: Subjects 54 Months After Booster Dose
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Started | 50 | 108 | 56
Completed | 50 | 108 | 56
Not Completed | 0 | 0 | 0
Period: Subjects 66 Months After Booster Dose
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Started | 48 | 104 | 53
Completed | 48 | 104 | 53
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group | Total
Number analyzed (Participants) | 58 | 123 | 57 | 238
Age, Continuous [Mean (Standard Deviation); unit: Months] — Baseline characteristics for Menitorix/Pediarix Group and Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group are given for subjects included in the Month 18 follow-up timepoint.
  For Infanrix Hexa/Meningitec Group, baseline characteristics are given for all subjects included in the Month 30 follow-up timepoint, as most subjects were eliminated from the Month 18 timepoint in this group.
  Months | 31.3 (0.54) | 31.4 (0.64) | 31.5 (0.87) | 31.4 (0.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics for Menitorix/Pediarix Group and Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group are given for subjects included in the Month 18 follow-up timepoint.
  For Infanrix Hexa/Meningitec Group, baseline characteristics are given for all subjects included in the Month 30 follow-up timepoint, as most subjects were eliminated from the Month 18 timepoint in this group.
  Participants
    Female | 27 | 55 | 27 | 109
    Male | 31 | 68 | 30 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Equal to or Above Cut-off Value of 1:8
Description: The cut-off value for the rSBA-MenC titers was equal to or above 1:8.
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after booster dose (day 0)
Population: Analysis was performed on the According-to-Protocol Cohort for antibody persistence, which included all subjects with evaluable data at each timepoint and who participated in the primary study (NCT00352963) and booster study (NCT00323050).
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 50 | 110 | 52
subjects
  Month 18 (N= 45; 96; 0) | 44 | 93 | 0
  Month 30 (N= 48; 101; 45) | 39 | 96 | 31
  Month 42 (N= 50; 110; 52) | 39 | 106 | 33
  Month 54 (N= 49; 106; 51) | 38 | 103 | 33
  Month 66 (N= 46; 101; 46) | 38 | 95 | 28

2. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Equal to or Above Cut-off Value of 1:32
Description: The cut-off value for the rSBA-MenC titers was equal to or above 1:32.
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 50 | 110 | 52
subjects
  Month 18 (N= 45; 96; 0) | 40 | 93 | 0
  Month 30 (N= 48; 101; 45) | 36 | 94 | 25
  Month 42 (N= 50; 110; 52) | 38 | 100 | 30
  Month 54 (N= 49; 106; 51) | 37 | 100 | 29
  Month 66 (N= 46; 101; 46) | 37 | 88 | 25

3. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titers Equal to or Above Cut-off Value of 1:128
Description: The cut-off value for the rSBA-MenC titers was equal to or above 1:128.
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 50 | 110 | 52
subjects
  Month 18 (N= 45; 96; 0) | 27 | 82 | 0
  Month 30 (N= 48; 101; 45) | 27 | 80 | 12
  Month 42 (N= 50; 110; 52) | 30 | 89 | 13
  Month 54 (N= 49; 106; 51) | 27 | 86 | 15
  Month 66 (N= 46; 101; 46) | 28 | 69 | 18

4. Primary Outcome: rSBA-MenC Titers
Description: Titers are expressed as Geometric Mean Titers (GMTs).
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after booster dose (day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 50 | 110 | 52
titer
  Month 18 (N= 45; 96; 0) | 221.5 [137.2 to 357.7] | 801.1 [570.3 to 1125.3] | 0 [0 to 0]
  Month 30 (N= 48; 101; 45) | 109.1 [61.9 to 192.3] | 441.7 [309.4 to 630.6] | 40.3 [21.9 to 74.1]
  Month 42 (N= 50; 110; 52) | 98.9 [56.7 to 172.5] | 409.8 [297.7 to 564.2] | 36.1 [20.4 to 63.8]
  Month 54 (N= 49; 106; 51) | 90.4 [52.8 to 154.8] | 344.6 [255.9 to 463.9] | 36.7 [21.1 to 64.0]
  Month 66 (N= 46; 101; 46) | 121.5 [71.0 to 207.9] | 227.6 [160.2 to 323.3] | 42.7 [22.3 to 81.8]

5. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Concentrations Equal to or Above Cut-off Value of 0.15 µg/mL (Microgram Per Milliliter)
Description: The cut-off value was an anti-PRP concentration equal to or above 0.15 µg/mL (microgram per milliliter).
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
subjects
  Month 18 (N= 56; 122; 3) | 56 | 121 | 3
  Month 30 (N= 53; 113; 53) | 53 | 112 | 53
  Month 42 (N= 50; 110; 51) | 50 | 109 | 51
  Month 54 (N= 49; 106; 52) | 49 | 105 | 52
  Month 66 (N= 47; 101; 47) | 47 | 101 | 46

6. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Concentrations Equal to or Above Cut-off Value of 1.0 µg/mL (Microgram Per Milliliter)
Description: The cut-off value was an anti-PRP concentration equal to or above 1.0 µg/mL (microgram per milliliter).
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
subjects
  Month 18 (N= 56; 122; 3) | 44 | 112 | 3
  Month 30 (N= 53; 113; 53) | 36 | 98 | 40
  Month 42 (N= 50; 110; 51) | 33 | 91 | 34
  Month 54 (N= 49; 106; 52) | 27 | 86 | 35
  Month 66 (N= 47; 101; 47) | 26 | 84 | 26

7. Primary Outcome: Anti-PRP Concentrations
Description: Concentrations are expressed as Geometric Mean Concentrations (GMCs) in µg/mL (microgram per milliliter).
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL (microgram per milliliter)
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
µg/mL (microgram per milliliter)
  Month 18 (N= 56; 122; 3) | 2.921 [2.150 to 3.968] | 5.450 [4.390 to 6.766] | 2.547 [0.390 to 16.651]
  Month 30 (N= 53; 113; 53) | 1.914 [1.383 to 2.648] | 3.524 [2.813 to 4.415] | 2.224 [1.578 to 3.133]
  Month 42 (N= 50; 110; 51) | 1.735 [1.243 to 2.423] | 2.986 [2.395 to 3.722] | 2.005 [1.365 to 2.946]
  Month 54 (N= 49; 106; 52) | 1.552 [1.154 to 2.087] | 2.688 [2.149 to 3.361] | 1.799 [1.267 to 2.555]
  Month 66 (N= 47; 101; 47) | 1.602 [1.107 to 2.320] | 2.625 [2.113 to 3.261] | 1.763 [1.170 to 2.657]

8. Primary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Concentrations Equal to or Above Cut-off Value of 0.3 µg/mL (Microgram Per Milliliter)
Description: The cut-off value was an anti-PSC concentration equal to or above 0.3 µg/mL (microgram per milliliter).
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
subjects
  Month 18 (N= 56; 122; 0) | 38 | 100 | 0
  Month 30 (N= 52; 108; 53) | 19 | 58 | 19
  Month 42 (N= 49; 107; 52) | 17 | 52 | 17
  Month 54 (N= 46; 105; 52) | 14 | 52 | 17
  Month 66 (45; 99; 45) | 12 | 34 | 11

9. Primary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Concentrations Equal to or Above Cut-off Value of 2.0 µg/mL (Microgram Per Milliliter)
Description: The cut-off value was an anti-PSC concentration equal to or above 2.0 µg/mL (microgram per milliliter).
  0 has been put as an arbitrary value for Month 18 in the Infanrix Hexa/Meningitec Group, as it was not addressed for reasons explained in the participant flow section.
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
subjects
  Month 18 (N= 56; 122; 0) | 1 | 31 | 0
  Month 30 (N= 52; 108; 53) | 1 | 18 | 3
  Month 42 (N= 49; 107; 52) | 0 | 14 | 2
  Month 54 (N= 46; 105; 52) | 1 | 10 | 1
  Month 66 (N= 45; 99; 45) | 0 | 8 | 0

10. Primary Outcome: Anti-PSC Concentrations
Description: Concentrations for anti-PSC antibody were expressed as GMCs.
Time Frame: 18, 30, 42, 54 and 66 months after the booster dose (day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL (microgram per milliliter)
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 56 | 122 | 53
µg/mL (microgram per milliliter)
  Month 18 (N= 56; 122; 0) | 0.50 [0.39 to 0.64] | 1.01 [0.80 to 1.29] | 0 [0 to 0]
  Month 30 (N= 52; 108; 53) | 0.26 [0.21 to 0.33] | 0.47 [0.37 to 0.61] | 0.30 [0.23 to 0.39]
  Month 42 (N= 49; 107; 52) | 0.25 [0.20 to 0.31] | 0.40 [0.32 to 0.51] | 0.28 [0.21 to 0.37]
  Month 54 (N= 46; 105; 52) | 0.24 [0.19 to 0.30] | 0.36 [0.29 to 0.45] | 0.26 [0.20 to 0.32]
  Month 66 (N= 45; 99; 45) | 0.22 [0.18 to 0.27] | 0.29 [0.23 to 0.36] | 0.22 [0.18 to 0.28]

11. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Serious adverse events assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From last study contact of the booster study (NCT00323050) to Month 66 after booster dose (day 0)
Population: Analysis was performed on the Total Cohort, which included all vaccinated subjects in the booster study (NC00323050) and who came back during the follow-up.
Measure: Number; unit: subjects
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Number analyzed (Participants) | 58 | 123 | 57
subjects | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the last contact of the booster study (NCT00323050) until Month 66 after the booster dose (day 0).
Description: For serious adverse events the amount of subjects at risk has been put as the maximum amount of subjects which have come back for this follow-up study. Other adverse events were not assessed.
Arm/Group | Menitorix/Pediarix Group | Infanrix Hexa (or IPV/Hib)/NeisVac-C/Engerix-B/Menitorix Group | Infanrix Hexa/Meningitec Group
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/123 | 0/57
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.